CLINICAL TRIAL: NCT07193472
Title: Analgesic Efficacy of Serratus Intercostal Plane Block Versus Port Infiltration in Laparoscopic Cholecystectomy: Randomised Clinical Trial
Brief Title: Serratus Intercostal Plane Block Versus Port Infiltration in Laparoscopic Cholecystectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital del Rio Hortega (Other)
Responsible Party: Principal Investigator, María Teresa Fernandez, MD, principal investigator, Hospital del Rio Hortega
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PI-25- 298-H; PI-25- 298-H (Other: RIO HORTEGA UNIVERSITY HOSPITAL)
Record Dates: First submitted 2025-06-24; First posted 2025-09-25 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Masking Description: both groups are masked about the receiving analgesia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- port infiltration (Other): patients receiving port infiltration as analgesia
  Interventions: Procedure: serratus intercostal plane block as analgesic technique

INTERVENTIONS:
Procedure: serratus intercostal plane block as analgesic technique — the SIPB will be applied after starting surgery and before general anaesthesia

SUMMARY:
Most patients undergoing laparoscopic cholecystectomy (LC) experience moderate to severe pain in the first 24 hours after surgery. Port infiltration is the usual analgesic method while serratus-intercostal plane blockade (SIPB) has shown its efficacy in open cholecystectomy pain control. The aim of the present study was to compare the efficacy of both techniques in pain control.

OBJECTIVE The prospective randomised study has the working hypothesis is based on evaluating whether serratus-intercostal block (modified BRILMA) is equal or superior to laparoscopic port infiltration (PI) in terms of quality of postoperative recovery and pain control.

Secondary objectives of the study will be to assess the absence of adverse effects.

MATERIAL AND METHODS the investigators present a low-intervention clinical trial. The sample will be composed of 128 patients divided into two groups according to the analgesic technique (serratus-intercostal and port infiltration), following a 1:1 randomisation, consecutively until the sample size is reached and fulfilling the following criteria: signature of informed consent, over 18 years of age, ASA I-III, undergoing laparoscopic cholecystectomy.

Intraoperatively, patients will receive standard monitoring and induction. Analgesia will consist of a multimodal strategy (8 mg dexamethasone, 1 g paracetamol and 50 mg dexketoprofen pre-incisionally, intraoperative fentanyl on demand and the corresponding regional technique).

In the postoperative period, the main variable to be evaluated in forms designed for this purpose will be the difference in pain assessed by means of an numeric rating scale (NRS scale) and the quality of recovery will be measured by means of the modified Postoperative Quality of Recovery Score (QoR-15 ) recovery scale (15 responses).

DETAILED DESCRIPTION:
Background

Postoperative pain remains a significant concern following laparoscopic cholecystectomy (LC), with most patients experiencing moderate to severe pain within the first 24 hours. Traditionally, port-site infiltration (PI) with local anesthetics is employed for analgesia. However, the serratus-intercostal plane block (SIPB), also known as the modified BRILMA block, has demonstrated efficacy in pain management for open cholecystectomy. Its role in LC remains to be clarified.

Objective

The primary objective of this prospective randomised study is to evaluate whether SIPB (modified BRILMA block) provides equivalent or superior postoperative analgesia and quality of recovery compared to port-site infiltration in patients undergoing LC.

Secondary objective: To assess the incidence of adverse effects related to each analgesic technique.

Methods

This study is designed as a low-intervention, prospective, randomized clinical trial. A total of 128 adult patients (ASA I-III) scheduled for elective laparoscopic cholecystectomy will be randomly allocated (1:1) to receive either serratus-intercostal plane block or laparoscopic port infiltration for perioperative analgesia. Randomization will be performed consecutively until the target sample size is reached.

Inclusion Criteria:

Age ≥ 18 years

ASA physical status I-III

Informed consent provided

Exclusion Criteria:

(Coagulopaty, allergy to local anaesthetic, history of chronic pain)

Intraoperative Management:

All patients will receive standardized general anesthesia and multimodal analgesia comprising:

8 mg dexamethasone

1 g paracetamol

50 mg dexketoprofen (administered pre-incisionally)

Fentanyl as needed during surgery

Assigned regional analgesic technique (SIPB or PI)

Postoperative Evaluation:

Primary Outcome Measures:

Pain intensity using the Numerical Rating Scale (NRS) at predefined intervals

Quality of recovery assessed via the modified QoR-15 questionnaire

Secondary Outcome Measure:Incidence of adverse events or complications related to the analgesic techniques

SIPB group: receive The Serratus intercostal plane block as analgesic technique after induction. With the patient lying in supine position, the local anaesthetic is administered in the plane under Serratus muscle at the 8th rib level Infiltration group: in this group the surgeons administered local anaesthetic after inserting the trocar.

Conclusion (anticipated)

This trial aims to determine whether SIPB offers superior analgesic efficacy and recovery quality compared to standard port infiltration in LC, potentially informing improved postoperative pain protocols.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II-III
* laparoscopic cholecystectomy

Exclusion Criteria:

* Alergy to used drugs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
efectiveness of analgesia (SIPB versus IP) | one year
  The working hypothesis is based on evaluating whether serratus-intercostal block (modified BRILMA) is equal or superior to laparoscopic port infiltration (PI) in terms of quality of postoperative recovery (QoR15) and pain control (NRS) 0-10

SECONDARY OUTCOMES:
side efects | one year
  assesment of side efects
Postoperative pain control | One year
  Pain developed for patients after surgery first 24 h . nRS 0-10
Postoperative recovery | One year
  Intake, rest at night, walking…assessed with QoR15 0- 150

CONTACTS AND LOCATIONS:
Overall Officials: Maria Teresa Fernandez, MD, Principal Investigator — Hospital del Rio Hortega
Locations (1):
- Fernandez, Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-05-25): https://cdn.clinicaltrials.gov/large-docs/72/NCT07193472/ICF_000.pdf